CLINICAL TRIAL: NCT04688242
Title: A Randomized, Phase 2 Study of Anal Dilatation Plus Probiotics Before Ileostomy Reduction for Low Anterior Resection Syndrome After Sphincter-preserving Proctectomy
Brief Title: Anal Dilatation Plus Probiotics Before Ileostomy Reduction for Low Anterior Resection Syndrome
Acronym: PILLARS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020ZSLYEC-187
Record Dates: First submitted 2020-12-13; First posted 2020-12-29 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2021-12

CONDITIONS: Low Anterior Resection Syndrome
Keywords: rectal cancer; temporary ileostomy; low anterior resection syndrome; anal dilatation; gut microbiota
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients were randomized to the treatment group (anal dilatation plus probiotics) or the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Anal dilatation plus probiotics per anus Q3D, starting from 2 weeks after proctectomy until reduction of ileostomy.
  Interventions: Other: Anal dilatation per anus; Drug: administration of probiotics (Clostridium butyricum TO-A; Bacillus mesentericus TO-A; Streptococcus faecalisT-110) per anus
- Control Arm (No Intervention): No anal dilatation or probiotics per anus was allowed, from 2 weeks after proctectomy until reduction of ileostomy.

INTERVENTIONS:
Other: Anal dilatation per anus — Digital anal dilatation through anastomosis, with concomitant administration of probiotics per anus
  Arms: Treatment Arm
Drug: administration of probiotics (Clostridium butyricum TO-A; Bacillus mesentericus TO-A; Streptococcus faecalisT-110) per anus — Digital anal dilatation through anastomosis, with concomitant administration of probiotics per anus
  Arms: Treatment Arm

SUMMARY:
This is randomized, phase 2 trial in patients with rectal cancer undergoing sphincter-preserving proctectomy and temporary ileostomy, to explore the effects of anal dilatation plus probiotics administered per anus before ileostomy reduction in relieving postoperative bowel dysfunction known as low anterior resection syndrome (LARS).

DETAILED DESCRIPTION:
Approximately 60-90% of patients undergoing sphincter-sparing proctectomy complain of postoperative bowel dysfunction including incontinence, frequency, clustering, and urgency, collectively known as low anterior resection syndrome (LARS). Literatures and our previous data have demonstrated that diverting ileostomy is an independent risk factor for major LARS. This is a randomized, phase 2 trial in patients with rectal cancer who underwent sphincter-preserving proctectomy and ileostomy. This study will explore the effects of anal dilatation plus probiotics administered per anus in relieving the symptoms of LARS.

ELIGIBILITY:
Inclusion Criteria:

1. A voluntarily signed and dated informed consent form;
2. ECOG Performance status is 0 or 1;
3. Age at enrollment is of 18 to 80 years old.;
4. R0 sphincter-preserving proctectomy and temporary ileostomy for rectal cancer;
5. The distance from anastomosis to anal verge is ≤7cm;
6. Both the anastomosis and the ileostomy is intact at 2 weeks follow-up after proctectomy;
7. Baseline LARS score before proctectomy is <30;
8. The preoperatively predicted LARS (POLARS) score after proctectomy is ≥28.

Exclusion Criteria:

1. R1/R2 resection or untreated metastases;
2. Any synchronous or metachronous malignancies, except for cancers that have received curative treatment and have not recurred for more than 5 years, or carcinoma in situ that have been cured by appropriate treatment;
3. Severe morbidity with life expectancy less than 2 years;
4. Any toxicity of CTCAE grade 2 or above due to previous treatment that have not resolved, except for anemia, alopecia, skin pigmentation;
5. Anastomotic leak within 2 weeks after proctectomy, suspected by clinical symptoms, digital rectal examination, or imaging;
6. Complications of the ileostomy within 2 weeks after proctectomy, leading to premature takedown of the stoma (within 2 months after surgery);
7. Any medical condition that may affect the safety and compliance of the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Major LARS at 1 years after proctectomy | At 1 years after proctectomy
  Proportion of patients with Low anterior resection syndrome (LARS) score ≥30. LARS score is a tool consisting of five items, which are as follows: incontinence due to flatus (score range from 0 to 7), incontinence due to liquid stools (score range from 0 to 3), frequency of bowel movements (score range from 0 to 5), clustering (score range from 0 to 11) and urgency (score range from 0 to 16). The severity of each item is calculated on a scale ranging from 0 to 42, with a score of 0-20 (no LARS), 21-29 (minor LARS) and 30-42 (major LARS).

SECONDARY OUTCOMES:
LARS score at 1 years after proctectomy | At 1 years after proctectomy
  Low anterior resection syndrome (LARS) score is a tool consisting of five items, which are as follows: incontinence due to flatus (score range from 0 to 7), incontinence due to liquid stools (score range from 0 to 3), frequency of bowel movements (score range from 0 to 5), clustering (score range from 0 to 11) and urgency (score range from 0 to 16). The severity of each item is calculated on a scale ranging from 0 to 42, with a score of 0-20 (no LARS), 21-29 (minor LARS) and 30-42 (major LARS).
Quality of life assessed using the EORTC Quality of Life questionnaire (QLQ)-C30 at 1 years after proctectomy | At 1 years after proctectomy
  The European Organisation for Research and Treatment of Cancer (EORTC) developed and validated a 30-item core questionnaire (QLQ-C30) reflecting global QoL in cancer patients. QLQ-C30 comprises five functional scales, three symptom scales, a global health scale/ a quality of life scale, and six single items. All the scales and single item measures range in score from 0-100. A high score represents a higher level of functioning, a high quality of life, and a greater degree of symptoms.
Quality of life assessed using the EORTC Quality of Life questionnaire (QLQ)-CR29 at 1 years after proctectomy | At 1 years after proctectomy
  QLQ-CR29 is developed by The European Organisation for Research and Treatment of Cancer (EORTC). It is a validated supplement to the QLQ-C30 specifically designed for assessment of quality of life in colorectal cancer patients. QLQ-CR29 consists of four functional scales and eighteen single items. All the scales range from 0-100. A high score represents a higher level of functioning and a greater degree of symptoms.
MSKCC BFI Score at 1 years after proctectomy | At 1 years after proctectomy
  The Memorial Sloan-Kettering Cancer Centre Bowel Function Instrument (MSKCC BFI) score is a validated questionnaire for evaluation of bowel function after sphincter-preserving surgery. It comprises 18 items covering the frequency of various LARS symptoms and is divided into three sub-scales and four single items. It is scored on a 5-point Likert scale ranging from "always" to "never". The sub-scales scores are summarised as: A 6-item frequency sub-scale (6-30), a four-item dietary sub-scale (4-20), and a four-item urgency sub-scale (4-20). A global score can be calculated as the sum of the sub-scale scores. A total score (possible score range 18-90) can be calculated by adding all the item scores (sub-scale scores plus single item scores). A higher score indicates better bowel function.
Presence of stoma at 1 years after proctectomy | At 1 years after proctectomy
  Proportion of patients with a stoma due to failure to reduce, or a second stoma after ileostomy reduction is assessed by a professional doctor or nurse at 2 years after proctectomy.
Anastomotic complications within 1 years after proctectomy | Within 1 years after proctectomy
  Anastomotic complications is assessed by a professional doctor using Common Terminology Criteria for Adverse Events (CTCAE) classification.
Time for major LARS (≥30) returning to minor or no LARS (<30) after proctectomy | Within 1 years after proctectomy
  LARS score is assessed every 6 months after proctectomy, and the time for major LARS (≥30) returning to minor or no LARS (<30) is recorded. Low anterior resection syndrome (LARS) score is a tool consisting of five items, which are as follows: incontinence due to flatus (score range from 0 to 7), incontinence due to liquid stools (score range from 0 to 3), frequency of bowel movements (score range from 0 to 5), clustering (score range from 0 to 11) and urgency (score range from 0 to 16). The severity of each item is calculated on a scale ranging from 0 to 42, with a score of 0-20 (no LARS), 21-29 (minor LARS) and 30-42 (major LARS).
Other complications within 1 years after proctectomy | Within 1 years after proctectomy
  Other complications is assessed by a professional doctor using Common Terminology Criteria for Adverse Events (CTCAE) classification.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - the Fifth Affiliated Hospital, Sun Yat-Sen University, Zhuhai, Guangdong